CLINICAL TRIAL: NCT00795327
Title: The Canadian Study of the Use of Injectable Poly-L-Lactic Acid Dermal Implant for the Treatment of Hill and Valley Acne Scarring
Brief Title: Injectable POLY-L-Lactic Acid for Treatment of Hill and Valley Acne Scarring
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bausch Health Americas, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: POLYL_L_02508
Record Dates: First submitted 2008-11-20; First posted 2008-11-21 (Estimated); Last update posted 2019-11-20 (Actual); Status verified 2019-11

CONDITIONS: Acne Vulgaris
MeSH Terms: conditions — Acne Vulgaris

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): single arm study
  Interventions: Device: Sculptra (Poly-L-Lactic Acid Dermal Implant)

INTERVENTIONS:
Device: Sculptra (Poly-L-Lactic Acid Dermal Implant) — Drug Device study

SUMMARY:
Primary:

Evaluate the degree of correction attainable with Poly-L-Lactic Acid(Sculptra) for the correction of hill and valley acne scarring

Secondary:

Document types and incidence of device adverse events with Poly-L-Lactic Acid(Sculptra) therapy.

ELIGIBILITY:
Inclusion Criteria:

* Outpatient seeking therapy for correction of hill and valley acne scarring.
* Ability and willingness to understand and comply with requirements of the trial

Exclusion Criteria:

* The subject has active acne or chronic skin disease, inflammation or related conditions, such as infection, psoriasis and herpes zoster
* History of presence of keloid formation or hypertrophic scars
* History of procedures that precipitate an active dermal inflammatory or hyperplastic response (i.e., epilation or radiofrequency laser and chemical peeling procedures) within one month of study entry
* History of use of facial tissue augmenting therapy or aesthetic facial surgical therapy within six months prior to study entry
* Concomitant anticoagulant therapy, antiplatelet therapy or has any bleeding disorders
* History of unanticipated adverse reactions when treated with hyaluronic acid based products
* Any condition which in the opinion of the investigator makes the patient unable to complete the study per protocol (e.g., patients not likely to avoid other facial cosmetic treatments; patients not likely to stay in the study for its duration because of other commitments, concomitant conditions, or past history; patients anticipated to be unreliable, or patients who have a concomitant condition that may develop symptoms that might confuse or confound study treatments or assessments)
* History of or current cancerous or pre-cancerous lesions in the area to be treated
* Use of any investigational drugs or any other medical devices within 30 days of enrolment
* Use of any prohibited medication within a proscribed time period before entry
* Pregnancy
* Recent use of Accutane (patient should not be on Accutane for the last 6 months)
* History of allergic/anaphylactic reactions, including hypersensitivity to local anaesthetics (lidocaine)
* Recent history of trauma in the face (less that 1 year)
* Previous of Dermalive or Dermadeep

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2008-10; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
Physician Scar Improvement Scale (PSIS) | At each visit
Self-Assessed Scar Improvement Scale (SASIS). | At each visit

SECONDARY OUTCOMES:
Degree of subject satisfaction with treatment | At each Visit
Adverse events | At each visit

CONTACTS AND LOCATIONS:
Overall Officials: Mary Tzortzis, Study Chair — Sanofi-Aventis Canada Inc.
Locations (1):
- Sanofi-Aventis Administrative Office, Laval, Canada